CLINICAL TRIAL: NCT05605249
Title: Remotely Prescribed and Monitored Home-based Gait-and-balance Therapeutic Exergaming Using Augmented Reality (AR) Glasses: Protocol for a Clinical Feasibility Study in People With Parkinson's Disease
Brief Title: Remotely Prescribed and Monitored Home-based Gait-and-balance Augmented Reality Exergaming for People With Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: Strolll, Ltd (Unknown)
Responsible Party: Principal Investigator, dr. Daphne J. Geerse, Principal Investigator, VU University of Amsterdam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL82441.100.22
Record Dates: First submitted 2022-09-30; First posted 2022-11-04 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Cue X; Augmented reality; Gait and balance exercise program; Clinical feasibility study
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The study consists of four visits to the gait laboratory and four contact moments by telephone divided over 13 weeks. In between visits 1 and 2 (period of 6 weeks), participants do not receive any training or instructions and will carry out their activities as normal. In between laboratory visits 2 and 4, participants will use Cue X to train their gait and balance with gamified AR gait-and-balance exercises in their own home environment as intervention above usual care (6 weeks for a minimum of 30 minutes per day and 5 days a week to comply with World Health Organization [2020] movement guidelines). Two different state-of-the-art AR headsets will be used for Cue X training, namely Microsoft's HoloLens 2 and Magic Leap's 2 headsets, randomized over participants using covariate adaptive randomization with age, gender and disease duration as covariates. Half of the participants will train with HoloLens 2 and the other half with Magic Leap 2.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cue X (Experimental): All participants will train with Cue X gamified AR gait-and-balance-exercises in their home environment for 6 weeks. Participants are invited to use Cue X minimally 5 times a week for 30 minutes total, but preferably on a daily basis. The exact exercises, exercise duration and difficulty level will be prescribed by a movement expert and will be evaluated and adjusted every week in telephone calls or during one of the laboratory assessment.
  Half of the participants will train with HoloLens 2 and the other half with Magic Leap 2.
  Interventions: Device: Cue X

INTERVENTIONS:
Device: Cue X — The Cue X movement training module includes several games that can be performed in someone's home environment. The games are designed based on known physiotherapy guidelines and evidence for improving motor symptoms for people with PD and delivered in AR. Some of the games also have integrated cueing to allow people with more severe mobility impairments to participate. Feedback of performance can be given using the movement data of the AR headsets.

SUMMARY:
Despite optimal treatment with medication, people with Parkinson's disease (PD) still experience symptoms and secondary complications. Physiotherapy has long been recognized as one of the leading treatments in PD for slowing progression of the disease and retaining a higher quality of life for longer. Physiotherapy includes, among other things, training motor functions e.g., gait, balance and strength training and encourages physical activity. Exercise is an important part of healthy living for everyone, but for people with PD, exercise is medicine. Studies even suggest that exercise may slow down disease progression. Another way of improving PD motor symptoms, such as festination and freezing of gait (FOG), in a more direct way is by sensory cueing. Cueing is defined as the application of spatial or temporal external stimuli to help initiate, or facilitate gait, and can be presented as acoustic, visual, or tactile stimuli. It has been well known for many years that sensory cueing is effective and there has been extensive research on the topic.

Cue X is a new product developed by Strolll Limited (www.strolll.co) that applies the existing proven principles of exercise and sensory cueing for PD onto augmented-reality (AR) headsets implemented in two modules: movement training and movement assistance. The movement training module is designed to train gait and balance in a gamified manner to maximize training compliance. With this clinical feasibility study, the investigators want to examine the feasibility and potential efficacy of the Cue X movement training module to train gait and balance of people with PD in their home environment.

DETAILED DESCRIPTION:
The primary objective of this clinical feasibility study in people with PD is to evaluate the feasibility and potential efficacy of home-based gamified AR gait-and-balance exercises with Cue X. Secondary objectives of this study are to validate the gait-modifying effects of Cue X AR cueing and to quantify the test-retest reliability and concurrent validity of (clinical) outcome measures of gait and balance, as derived from AR headset data.

With these primary and secondary objectives, the study will give insight into 1) the feasibility and potential efficacy of Cue X for home-based gamified AR gait-and-balance exercises, 2) the most effective type of AR cueing and 3) the best parameters for feedback, reporting and sample-size calculations for a subsequent effect study with Cue X. Furthermore, the study will inform about the best AR headset for these purposes.

ELIGIBILITY:
Inclusion Criteria:

* Have command of the Dutch language
* Diagnosed with PD according to the UK PD Brain Bank criteria (stages 2-4 on the Hoehn and Yahr scale)
* Bothersome gait or balance impairments (i.e., negatively affecting their ability to perform their usual daily activities)

Exclusion Criteria:

* Inability to comply with the protocol, i.e. additional neurological diseases and/or orthopaedic problems seriously interfering with gait function, insufficient physical capacity or cognitive/communicative inability (as observed by the researcher or clinician) to understand instructions and participate in the tests
* Visual or hearing impairments (after corrective aids)
* Severe visual hallucinations or illusions
* Inability to walk independently for 30 minutes
* No stable dosage of medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) [Usability] | After 6-week training
  A 10-item questionnaire to measure usability of the Cue X training module, answered on a 5 point Likert scale (1 strongly disagree - 5 strongly agree). Minimum - maximum score: 10 - 50. Higher scores imply better usability of the Cue X software.
Number of adverse events [safety] | During 6-week training
  To measure safety of the Cue X training module
Side effects as reported by participants [safety] | During 6-week training
  To measure safety of the Cue X training module
Adherence to the training programme | During 6-week training
  Actual exercise time as a percentage of prescribed exercise time. The prescribed exercise time is 30 minutes, 5 days a week.
Patient-reported outcome measures (PROMs) | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  An example is quality of life as measured by the Parkinson's Disease Questionnaire (PDQ-39). This questionnaire assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living, among which quality of life. Higher scores on one of the dimensions indicate worse well-being on that specific dimension.
Patient-reported experience measures (PREMs) | After 6-week training
  Perceived effectiveness of the Cue X training programme through Likert scale reporting and semi-structured interview questions during weekly phone calls and a post-intervention interview.
Mini Balance Evaluation Systems Test (Mini-BESTest) [Gait-and-balance outcome measures] | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  To measure balance and postural control. Minimum - maximum score: 0 - 28. Higher scores indicate better balance and postural control.
Timed Up-and-Go test (TUG) [Gait-and-balance outcome measures] | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  To measure functional gait. Higher scores indicate worse functional gait.
Lindop Parkinson's Physiotherapy Assessment Scale (LPPAS) [Gait-and-balance outcome measures] | Change between pre-, mid- and post-training measure (over 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  To measure gait mobility. Higher scores indicate better gait mobility. Minimum - maximum score: 0 - 18
Targeted walking-related fall-risk assessment as measured by the Interactive Walkway | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  Targeted walking-related fall-risk assessment based on outcome measures of walking adaptability as determined with the Interactive Walkway (obstacle avoidance margins and success rates and stepping accuracy and walking speed during goal-directed stepping)

SECONDARY OUTCOMES:
Five Times Sit to Stand Test (FTSTS) | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  To measure lower extremity strength [standard clinical tests and questionnaires]. Higher scores indicate worse lower extremity strength.
New Freezing of Gait Questionnaire (NFOGQ) | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  To measure freezing of gait severity [standard clinical tests and questionnaires]. Higher scores indicate the severity and the burden of freezing of gait in daily life is worse. Minimum - maximum score: 0 - 28.
Movement Disorders Society Unified Parkinson Disease Rating Scale (UPDRS) | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  To measure overall PD severity [standard clinical tests and questionnaires]. The UPDRS consists of three segments: I) Mentation, Behavior and Mood, II) Activities of Daily Living, and III) Motor Examination. Higher scores on these segments and higher total scores indicate more severe PD symptoms.
Activities-Specific Balance Confidence Scale (ABC) | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  To measure balance confidence [standard clinical tests and questionnaires]. Minimum - maximum score: 0 - 1600. Higher scores indicate more confidence in performing daily activities without losing balance.
Falls Efficacy Scale International (FES-I) | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  To measure fear of falling [standard clinical tests and questionnaires]. Minimum - maximum score: 16 - 64. Higher scores indicate that the participant is more concerned about falling.
Physical Activity Scale for the Elderly (PASE) | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  To measure physical activity [standard clinical tests and questionnaires]. Higher scores indicate greater physical activity.
Gait speed [Gait-modifying ability and data quality] | Change between pre-, mid- and post-training measure (over 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  Spatiotemporal gait parameters (speed, cadence, step length, step time) derived from Interactive Walkway and AR headsets during the 8-meter walking test (with or without visual/auditory cues) and standard clinical tests of gait and balance derived from AR headsets and stopwatch scores
Cadence [Gait-modifying ability and data quality] | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  Spatiotemporal gait parameters (speed, cadence, step length, step time) derived from Interactive Walkway and AR headsets during the 8-meter walking test (with or without visual/auditory cues) and standard clinical tests of gait and balance derived from AR headsets and stopwatch scores
Step length [Gait-modifying ability and data quality] | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  Spatiotemporal gait parameters (speed, cadence, step length, step time) derived from Interactive Walkway and AR headsets during the 8-meter walking test (with or without visual/auditory cues) and standard clinical tests of gait and balance derived from AR headsets and stopwatch scores
Step time [Gait-modifying ability and data quality] | Change between pre-, mid- and post-training measure (over a period of 12 weeks, which includes 6 weeks waiting list and 6-week intervention)
  Spatiotemporal gait parameters (speed, cadence, step length, step time) derived from Interactive Walkway and AR headsets during the 8-meter walking test (with or without visual/auditory cues) and standard clinical tests of gait and balance derived from AR headsets and stopwatch scores

CONTACTS AND LOCATIONS:
Overall Officials: Melvyn Roerdink, PhD, Study Director — VU University of Amsterdam
Locations (1):
- Vrije Universiteit Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
This study is part of a collaboration between the Vrije Universiteit Amsterdam and Strolll, the manufacturer of Cue X. Movement- and/or environmental data from the headsets and gold standards and information on adherence (e.g., tasks performed, hours spend on games) of this study will be shared anonymously with Strolll to be used for the further development of Cue X.
  Anonymized research data will be published along with articles as supplemental material or will be made available in a repository.

REFERENCES:
- [Background] Hardeman LES, Geerse DJ, Hoogendoorn EM, Nonnekes J, Roerdink M. Remotely prescribed and monitored home-based gait-and-balance therapeutic exergaming using augmented reality (AR) glasses: protocol for a clinical feasibility study in people with Parkinson's disease. Pilot Feasibility Stud. 2024 Mar 27;10(1):54. doi: 10.1186/s40814-024-01480-w. PMID 38539250
- [Background] Hardeman LES, Geerse DJ, Hoogendoorn EM, Nonnekes J, Roerdink M. Remotely prescribed, monitored, and tailored home-based gait-and-balance exergaming using augmented reality glasses: a clinical feasibility study in people with Parkinson's disease. Front Neurol. 2024 May 30;15:1373740. doi: 10.3389/fneur.2024.1373740. eCollection 2024. PMID 38872812